CLINICAL TRIAL: NCT03428347
Title: An Open, Dose Escalation Safety and Pharmacokinetics Study of the Medicine for Ebola Fever Emergency Prevention Based on Monoclonal Recombinant Antibodies With a Single Application in 3 Groups of Healthy Volunteers
Brief Title: An Open Study of the Safety and Pharmacokinetics of a Medicinal Product for Emergency Prevention of Ebola
Acronym: 03-AT-2017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Research Institute of Influenza, Sankt-Peterburg, Russian Federation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-AT-2017
Record Dates: First submitted 2018-01-25; First posted 2018-02-09 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Ebola; Ebola Virus Disease; Monoclonal antibody
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 1.4 mg/kg body weight
  Interventions: Biological: GamEMab
- Group 2 (Experimental): 7 mg/kg body weight
  Interventions: Biological: GamEMab
- Group 3 (Experimental): 14 mg/kg body weight
  Interventions: Biological: GamEMab

INTERVENTIONS:
Biological: GamEMab — drug for emergency prevention of Ebola based on recombinant monoclonal antibodies

SUMMARY:
This Phase I clinical trial was developed to study drug safety, tolerability, and pharmacokinetics of the medicine for Ebola fever emergency prevention based on monoclonal recombinant antibodies in single use in healthy volunteers with a dose escalation. A consecutive recruitment of people who signed the Informed Consent Form into three groups of volunteers with different drug doses is made according to the volunteers' screening results. The total number of volunteers receiving the drug will be not less then 25 people.The purpose of this study is to assess safety, tolerability, and pharmacokinetics of a medicine for Ebola fever emergency prevention based on monoclonal recombinant antibodies in a single dose in healthy volunteers.

DETAILED DESCRIPTION:
The results of the screening of volunteers who signed the informed consent Form, is a sequence set in three groups of volunteers with different doses of the drug, the total number of volunteers who received the drug will be at least 25 people.

Taking into account the fact that for the first time the drug is studied on people, initially five volunteers will be hospitalized. Their dose of the studied medicine will be 1.4 mg/kg of weight. After confirmation of safety based on observation results on the 60th day of the study, the investigation will continue with the participation of five more volunteers. Safety will be studied on these five volunteers with a single use of dose of 7 mg/kg of weight.

After an intermediate safety assessment on the 60th day, 15 more volunteers will be included in the study. They will get the medicine with the dose of 14 mg/kg of weight.

If necessary, understudies in an amount of not more than 4 people may be included. Volunteers are replaced before the injection of the medicine. If a volunteer got the medicine, he could not be replaced.

After evaluating the safety analyzes' intermediate results (blood test and blood chemistry, urinalysis, immunological safety, clinical evaluation of general health status) obtained on day 60 of the study, the Researcher, in agreement with the Ethics Committee, makes a decision to include the second group (five people) to study the drug at a dosage of 7 mg/kg of weight. After the evaluation of intermediate safety results on the 60th day of the study of volunteers from the second group, 15 more volunteers will be included in the study. After the intermediate evaluation of safety on the 60th day of study, 15 more volunteers will be included in the study and get the medicine in a dose of 14 mg/kg of weight. Wherein the third part of volunteers is planned to be included consistently: in the beginning 5 volunteers will be included and after the intermediate safety evaluation on the 28th day the rest 10 volunteers will be included in the study.

The safety and tolerability assessment will be based on the registration of adverse events during the study. Changes in instrumental (ECG) and laboratory indicators (blood test and blood chemistry, blood coagulation system indicators, urinalysis, immunological status), dynamics of vital signs (blood pressure, heart rate, body temperature) will be also evaluated.

Pharmacokinetic parameters will be calculated by a model-independent method. Immunological methods (ELISA) will be used for studying the level of specific antibodies and the duration of their circulation in the human body.

Sampling of biological material involves:

Urinalysis: at screening, before administration of the drug after 48 hours and on 7, 10, 14, 21, 28, 45, 60 and 90 days of the study; urine samples for a pregnancy test taken at screening and on the day of hospitalization (in addition to volunteers women).

to define security settings (General clinical and biochemical** blood tests, including a study of the coagulation system): at screening, before dosing, 48 hours, and 7, 10, 14, 21, 28, 45, 60 and 90 days of the study; immune status***- the drug, 7, 10, 14, 21, 28, 45, 60 and 90 days of the study; will also be determining the level of specific antibodies to the drug (with detection with the determination of class, subclass, immunoglobulins and assessment of their functional activity) is the drug, 7, 10, 14, 21, 28, 45, 60 and 90 days of the study; **biochemical blood analysis includes a determination of: total protein, urea, creatinine, aspartataminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin, glucose, cholesterol, creatine phosphokinase, CRP, concentration of electrolytes (sodium, potassium), coagulation include: PI+, INR, APTT, fibrinogen.

*** evaluation of the immunological status includes: determining the number and relative content of subpopulations of T - and b-lymphocytes (CD3, CD 4, CD 8, CD 16, CD19), phagocytic activity of white blood cells, immunoregulatory index, content of serum immunoglobulins major classes (A, M, G, E), circulating immuno complexes, the detection of antibodies to the mouse immunoglobulin, the content of anti-inflammatory cytokines (TNF-α, ИЛ1, IL-6, IFN-γ).

Blood samples for testing for hepatitis b and C, HIV and syphilis will be taken once at screening visit.

In addition there will be samples of whole blood for analysis of pharmacokinetic parameters: before drug administration, through 1, 4, 8, 24, 36, 48 and 96 hours after drug administration, and 7, 10, 14, 21, 28, 45, 60 and 90 days study.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 45 years;
* written informed consent;
* consent to use of effective contraception methods during the whole period of participation in the study; (using one of the following methods: abstinence, condoms (male or female with or without spermicide), diaphragm or cervical cap with a spermicidal tool, intrauterine device);
* body mass index (BMI) is 18.5 ≤ BMI ≤ 30;
* absence of acute infections/exacerbations of chronic at the time of participation in the study and for 7 days before initiation of therapy;
* absence of allergic disease severe disease (anaphylaxis, angioedema, polymorphic exudative eczema, serum sickness);
* no history of severe complications in a previous application of immunobiological preparations;
* lack of history, but also according to screening tests, pathology of the gastrointestinal tract, liver, kidneys, cardiovascular system, Central nervous system, musculoskeletal, urogenital and endocrine systems that can influence the evaluation of the results of the study;
* negative pregnancy test blood or urine (for women of childbearing age) not more than 24 hours before receiving the first dose of study drug;
* negative tests for HIV, hepatitis b and C, syphilis;
* negative urine test for drug traces;
* negative test for alcohol content in breath;
* absence of malignant blood diseases;
* absence of malignant tumors;
* negative allergological study on the epithelium and the proteins of the mouse.
* anti-mouse antibody titer less than 1:500;
* indicators of the General analysis of blood, biochemical analysis of blood total IgE at screening within the normal values.

  *( will be provided normal reference values of the laboratory performing the study)
* no history of previous vaccination against Ebola, including during clinical studies

Exclusion Criteria:

* volunteer participation in any other clinical trial within the last 90 days;
* respiratory symptoms in the last 3 days;
* treatment with steroids for the last 10 days (excluding preparations for intranasal administration and topical application);
* allergic reactions to proteins/epithelium of the mouse in history or about the results of laboratory studies on the screening, the titer of anti-mouse antibodies according to the study of 1:500 and more; introduction immunoglobulins or other blood products within the last 6 months;
* treatment with immunosuppressive drugs and/or immunomodulators within 6 months prior to the study;
* the use of other drugs based on murine monoclonal antibodies in history;
* regular past or current use of narcotic drugs;
* pregnancy or breast-feeding;
* systolic blood pressure less than 100 mm of mercury.St. or above 139 mm Hg.St; diastolic blood pressure less than 60 mm of mercury.St. or higher 90 mm. Hg.St.; heart rate less than 60 beats/min or more than 90 beats/min;
* aggravation of allergic diseases, the presence of anaphylactic reactions or angioedema in history;
* allergic reactions to the drug components;
* the presence of comorbid disease that may influence the assessment of the research results: active tuberculosis, chronic diseases of the liver and kidneys, expressed violations of function of thyroid gland and other endocrine system diseases (diabetes), severe diseases of the hematopoietic system, epilepsy and other diseases of the Central nervous system, myocardial infarction in anamnesis, myocarditis, endocarditis, pericarditis, ischemic heart disease, autoimmune disorders, severe chronic diseases that require hospital observation, and other diseases according to the researcher, will not allow the volunteer to participate in the study or may influence the research and/or its results (including the valuation of security);
* donating blood (450 ml blood or plasma, and more) in less than 2 months before the study;
* receiving history more than 5 units (0.25 l of ethanol) of alcohol per week;
* Smoking more than 10 cigarettes per day;
* planned hospitalization and/or surgical intervention during participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Adverse Events

SECONDARY OUTCOMES:
Number of Participants With Serious Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Serious Adverse Events
Number of Participants with Solicited Local and Systemic Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants with Solicited Local and Systemic Adverse Events
Pharmacokinetics Study | before drug administration, after 1, 4, 8, 24, 36 and 48 hours after drug administration, and 7, 10, 14, 21, 28, 45, 60 and 90 days study.
  Immunological methods will be used to study the level of specific antibodies and the duration of their circulation in the human body (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Lyoznov, MD, PhD, Principal Investigator — Research Institute of Influenza, Sankt-Peterburg, Russian Federation
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No